CLINICAL TRIAL: NCT05041010
Title: A Phase III, Double-blind, Randomized, Placebo-controlled, Multi-center Study to Assess the Efficacy and Safety of Nelonemdaz in Patients With Acute Ischemic Stroke
Brief Title: Rescues On Reperfusion Damage In Cerebral Infarction by Nelonemdaz
Acronym: RODIN
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: GNT Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Neu2000KWL-P03
Record Dates: First submitted 2021-09-02; First posted 2021-09-10 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2021-09

CONDITIONS: Ischemic Stroke
Keywords: Neu2000KWL; Neuroprotection; endovascular therapy; glutamate; free radical
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neu2000KWL (Experimental)
  Interventions: Drug: Neu2000KWL group
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo group

INTERVENTIONS:
Drug: Neu2000KWL group — 1st infusion of 750mg in patients receiving endovascular therapy within 12 hours following ischemic stroke onset followed by 9 consecutive infusions of 500 mg at intervals of 12 ± 1 hours, twice a day.
  Arms: Neu2000KWL
Drug: Placebo group — 1st infusion of the same volume of saline in patients receiving endovascular therapy within 12 hours following ischemic stroke onset followed by 9 consecutive infusions of same volume of saline at intervals of 12 ± 1 hours, twice a day
  Arms: Placebo

SUMMARY:
Efficacy and safety of Neu2000, a multi-target drug designed to prevent both NMDA receptor-mediated excitotoxicity and free radical toxicity, will be investigated in acute ischemic stroke patients receiving endovascular treatment to remove clot within 12 hours following stroke onset. Neu2000KWL will be administered before endovascular treatment.

DETAILED DESCRIPTION:
Neu2000 was designed as a multi-target neuroprotectant preventing both the NMDA receptor, a Ca2+ -permeable glutamate receptor, and free radicals, two major routes of brain cell death in stroke. Neu2000 is a moderate NR2B-selective NMDA receptor antagonist and spin trapping molecule (=free radical scavenger or antioxidant). Therapeutic potential of Neu2000 has been well demonstrated in four animal models of stroke with better efficacy and therapeutic time windows than either NMDA receptor antagonist or anti-oxidant advanced to clinical trials. In human phase I studies of 165 healthy subjects conducted in the United States and China, Neu2000KWL showed promising safety profiles without any serious adverse events up to a single intravenous infusion of 6000 mg that is far beyond the therapeutic target dose determined in animal models of transient ischemic stroke. Very recently, acute endovascular recanalization therapy has been introduced as the new standard care of care in acute ischemic stroke. The present study is aimed to examine efficacy and safety of Neu2000KWL in acute ischemic stroke patients receiving endovascular thrombectomy within 12 hours of stroke onset. This is a randomized trial, with placebo comparison, of comparing functional outcome at week 12 after 10 times of administration for five days.

ELIGIBILITY:
Inclusion Criteria:

The trial subjects should satisfy all the following criteria.

1. Adults≥19 years
2. Patients who can start endovascular therapy within 12 hours after the symptomatic onset of Ischemic stroke.
3. NIHSS on screening time point ≥ 8 points
4. Patients whose general condition was favorable enough to perform daily activities without the help of others one day prior to the ischemic stroke onset (a person with mRS 0 or 1)
5. Patients whose CTA or MRA confirmed internal carotid artery occlusion and M1 or M2 occlusion of the middle cerebral artery, that are the types of major cerebral artery occlusion that can cause acute cerebral infarction and are subject to endovascular therapy.
6. Patients with early ASPECTS point≥4 (Noncontrast brain cross-section CT or Brain cross-section MRI diffusion weighted imaging)
7. Patients who spontaneously submitted a written informed consent to participation on this clinical study.

Exclusion Criteria:

A patient who meets any one of the conditions below cannot participate in the Clinical trial.

1. Patients who meet the following exclusion criteria on imaging of endovascular therapy

   ① Patients whose occlusion location that can cause an acute ischemic stroke in the CTA (CT angiography) image meets under the following conditions: A. Occlusion of bilateral large artery B. Simultaneous infiltration of anterior and posterior circulation
2. Patients who have contraindication to contrast media for brain imaging.
3. Patients who are receiving renal replacement therapy such as dialysis due to acute or terminal nephropathy at screening point.
4. Patients who were diagnosed with cancer or received cancer therapy within 6 months at screening or have recurrent or transitional cancer.
5. Patients have high body temperature of 38oC or more and need antibiotic therapy due to medical opinion of infectious disease at screening.
6. Patients who are having pharmacotherapy due to liver diseases such as hepatic cirrhosis, etc. at screening point.
7. Patients who are pregnant or lactating. However, only a woman who has no possibility of pregnancy can participate in this clinical research.

   Woman with child-bearing potential can be defined as the woman who has not had the clear menopause or who has not had surgical treatment that makes pregnancy impossible.
8. Patients who have participated in other clinical trial within past 6 months at the screening time as a base. However, in case of participation of observatory experiment, the patient can participate in this clinical trial.
9. Patients who are determined unsuitable for participation in this clinical trial due to other reasons

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 496 (Estimated)
Dates: Start 2021-12-25 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
mRS score evaluated at 12 week after the first dose of drug (Nelonemdaz or Placebo). | week12

SECONDARY OUTCOMES:
Proportion of mRS 0-2 evaluated at week 5 and week 12 after the first dose of drug (Nelonemdaz or Placebo). | week5, week12
mRS score evaluated at week 5 after the first dose of investigational drug (Nelonemdaz or Placebo). | week5
Proportion of mRS 0 measured at week 5 and week 12 after the first dose of investigational drug (Nelonemdaz or Placebo). | week5, week12
Proportion of NIHSS 0-4 evaluated within 24 hours (Within 72 hours if weekend is included), 5 week, 12 week after the last injection of drug. (Evaluating 43 points for deaths) | 24hour(or 72hour), week5, week12
Volume of Ischemic stroke based on brain MRI diffusion weighted imaging within 24 hours and at week 12. (If MRI is not available, reading will be performed based on CT scan.) | 24hour, week12
Proportion of Barthel Index≥95 evaluated at week 5 and week 12 | week5, week12
Occurrence rate of Symptomatic intracranial hemorrhage (SICH) described and defined by this study occurring within 24 hours after the last injection | 24hour
  [Definition of Symptomatic intracranial hemorrhage (SICH)] In the case that brain imaging confirms intracranial hemorrhage with neurological deterioration. (NIHSS score≥4 points) neurological deterioration. (NIHSS score≥4 points)

OTHER OUTCOMES:
Proportion of adverse events and serious adverse events | day0~week12
All mortality rate until 12 weeks | day0~week12

CONTACTS AND LOCATIONS:
Overall Officials: Sun Uck Kwon, MD, PhD, Principal Investigator — Department of Neurology Asan Medical Center
Locations (24):
- South Korea (24):
  - Inje University Busan Paik Hospital, Busan
  - Dong-A University Hospital, Busan
  - Gyeongsang National University Hospital, Changwon
  - Chungbuk National University Hospital, Cheongju-si
  - Kyungpook National University Hospital, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - Daejeon Eulji Medical Center, Eulji University, Daejeon
  - Chosun University Hospital, Gwangju
  - Chonnam National University Hospital, Gwangju
  - Hallym University Dongtan Sacred Heart hospital, Hwaseong
  - Wonkwang University Hospital, Iksan
  - Gachon University Gil Medical Center, Incheon
  - Inha University Hospital, Incheon
  - Jeju National University Hospital, Jeju City
  - Jeonbuk National University Hospital, Jeonju
  - Seoul National University Bundang Hospital, Seongnam
  - Kyunghee University Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Ewha womans University Seoul Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Ulsan University Hospital, Ulsan
  - Yongin Severance Hospital, Yŏngin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lee JS, Kang HG, Ahn SH, Song TJ, Shin DI, Bae HJ, Kim CH, Heo SH, Cha JK, Lee YB, Kim EG, Park MS, Park HK, Kim J, Yu S, Mo H, Sohn SI, Kwon JH, Kim JG, Kim YS, Choi JC, Hwang YH, Jung KH, Kim SK, Seo WK, Seo JH, Yoo J, Chang JY, Park M, Lee JS, San An C, Gwag BJ, Choi DW, Kwon SU. Nelonemdaz and Patients With Acute Ischemic Stroke and Mechanical Reperfusion: The RODIN Randomized Clinical Trial. JAMA Netw Open. 2025 Jan 2;8(1):e2456535. doi: 10.1001/jamanetworkopen.2024.56535. PMID 39874036
- [Derived] Lee JS, Lee JS, Gwag BJ, Choi DW, An CS, Kang HG, Song TJ, Ahn SH, Kim CH, Shin DI, Kwon SU. The Rescue on Reperfusion Damage in Cerebral Infarction by Nelonemdaz (RODIN) Trial: Protocol for a Double-Blinded Clinical Trial of Nelonemdaz in Patients with Hyperacute Ischemic Stroke and Endovascular Thrombectomy. J Stroke. 2023 Jan;25(1):160-168. doi: 10.5853/jos.2022.02453. Epub 2023 Jan 31. PMID 36746385